CLINICAL TRIAL: NCT00289289
Title: Reducing Episodes by Septal Pacing Efficacy Confirmation Trial (RESPECT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 217
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation; Tachycardia, Supraventricular; Arrhythmia; Bradycardia
Keywords: Atrial Fibrillation; Atrial Tachyarrhythmia; Arrhythmia; Bradycardia; Cardiac Pacemaker; IPG Indication; Pacing
MeSH Terms: conditions — Atrial Fibrillation; Tachycardia, Supraventricular; Arrhythmias, Cardiac; Bradycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- On-Off (Active Comparator): Subjects have intervention pacing features turned On according to randomization assignment in the first crossover period then Off in the second period.
  Interventions: Device: Intervention Pacing Features
- Off-On (Active Comparator): Subjects have intervention pacing features turned Off according to the randomization assignment for the first crossover period and then On in the second period.
  Interventions: Device: Intervention Pacing Features
- Non-randomized (No Intervention): Subjects that did not have device recorded episodes of atrial tachycardia/atrial fibrillation during the 3 month observation period post-implant did not qualify for randomization but were continued to be followed in the study. There were no programming requirements and symptom activations were not collected.

INTERVENTIONS:
Device: Intervention Pacing Features — Intervention pacing features (atrial rate stabilization algorithm, atrial preference pacing algorithm, post mode switch overdrive pacing algorithm) in the pacemaker.
  Arms: Off-On; On-Off

SUMMARY:
The purpose of this study is to find out if specialized programs in the AT500 and EnRhythm pacemakers will reduce the number of irregular heartbeat in the upper chamber of the heart and reduce symptoms (such as shortness of breath, dizziness, and others).

DETAILED DESCRIPTION:
The purpose of the study was to confirm the AT500 intervention pacing effectiveness data previously seen in the ASPECT clinical trial and to gather additional data to understand the effectiveness of the intervention pacing features. Specifically, the goal of the trial is to demonstrate a reduction in frequency in symptomatic atrial tachycardia/atrial fibrillation recurrence with the intervention pacing features in patients with a pacing indication and a history of atrial tachyarrhythmias with atrial pacing leads located in the region of Bachmann's Bundle.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with fast and/or slow heartbeats who are in need of dual chamber pacing (pacing in both the atria and ventricles) as determined by their doctor.
* Subjects who have a history of occasional fast heartbeats originating from the upper heart chambers.
* Subjects who have experienced at least two symptomatic episodes of fast heartbeats three months prior to enrollment.
* Subjects that are expected to stay on the same heart medications during the length study.

Exclusion Criteria:

* Subjects who have permanent (chronic) or persistent (not self-terminating) atrial fibrillation (fast heartbeats originating from the upper heart chambers).
* Subjects who have atrial fibrillation due to a reversible cause, i.e. electrolyte imbalance.
* Subjects who are current or immediate implantable cardioverter defibrillator (ICD) recipients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2004-02; Primary Completion 2010-11 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RESPECT Team, Study Chair — Medtronic
Locations (38):
- United States (34):
  - Little Rock, Arkansas
  - Rancho Mirage, California
  - San Diego, California
  - Yuba City, California
  - Colorado Springs, Colorado
  - Jacksonville, Florida
  - Lakeland, Florida
  - Chicago, Illinois
  - Decatur, Illinois
  - Urbana, Illinois
  - Indianapolis, Indiana
  - Cedar Rapids, Iowa
  - Louisville, Kentucky
  - Owensboro, Kentucky
  - Takoma Park, Maryland
  - Springfield, Massachusetts
  - Minneapolis, Minnesota
  - Clifton, New Jersey
  - Morristown, New Jersey
  - Albuquerque, New Mexico
  - Mineola, New York
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Columbus, Ohio
  - Hershey, Pennsylvania
  - Spartanburg, South Carolina
  - Amarillo, Texas
  - Austin, Texas
  - Corpus Christi, Texas
  - Fort Worth, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Richmond, Virginia
  - Morgantown, West Virginia
- Canada (4):
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Kingston, Ontario
  - Sherbrooke, Quebec

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first study implant occurred on 13 February 2004 and the last study visit occurred on 10 November 2010
Pre-assignment Details: At the 3-month post-implant follow-up visit, all implanted subjects with documented Atrial tachycardia/Atrial fibrillation episode(s) during the 3-month observation period were eligible for randomization. Subjects with no documented Atrial tachycardia/Atrial fibrillation episodes were followed as part of the non-randomized group.
Groups:
- Non-Randomized Group: Subjects exiting prior to the 3-month randomization visit or subjects with no AT/AF burden during the 3-month observation period
Period: Overall Study
Arm/Group | On-Off | Off-On | Non-Randomized Group
Started | 132 | 124 | 144
Completed | 113 | 114 | 95
Not Completed | 19 | 10 | 49
Not completed — Withdrawal by Subject | 5 | 3 | 15
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Death | 4 | 2 | 5
Not completed — No implant attempted | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 6
Not completed — Non-study device implanted | 2 | 1 | 3
Not completed — Did not meet inclusion/exclusion | 0 | 0 | 6
Not completed — Other Exit Reason | 6 | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-Off | Off-On | Non-Randomized Group | Total
Number analyzed (Participants) | 132 | 124 | 144 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 30 | 27 | 82
  >=65 years | 107 | 94 | 117 | 318
Age Continuous [Mean (Standard Deviation); unit: years] | 73.0 (9.9) | 70.6 (9.3) | 72.4 (9.2) | 72.0 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 60 | 80 | 222
  Male | 50 | 64 | 64 | 178
Region of Enrollment [Number; unit: participants]
  United States | 125 | 118 | 139 | 382
  Canada | 7 | 6 | 5 | 18

OUTCOME MEASURES:

1. Primary Outcome: Rate of Symptomatic Atrial Tachycardia/Atrial Fibrillation Episodes Per Subject Per Month
Description: The frequency of symptomatic atrial tachycardia/atrial fibrillation (AT/AF) episodes as measured by the Patient Assistant and retrieved from save-to-disk information. For each subject and programming period (3-9 month period and 9-15 month period), the rate of symptomatic AT/AF episodes was computed by summing the total number of Patient Assistant activations during device recorded AT/AF episodes divided by months of device follow-up in each study period. Within each subject, the ON minus OFF difference in rate of symptomatic AT/AF was computed
Time Frame: 6-months (per Intervention)
Population: Patient Assistant data which contained markers for symptomatic atrial tachycardia or atrial fibrillation episodes obtained from save-to-disk data was required from both randomized follow-up periods (3-9 months and 9-15 months) for the subject to be included in the primary ITT analysis.
Measure: Mean (Standard Deviation); unit: Episodes per subject per month
Groups:
- Intervention Pacing Features Programmed ON: 6-month period subjects had the intervention pacing features programmed ON. For subjects randomized to the ON-OFF group, this was the 3-9 month post-implant period. For subjects randomized to the OFF-ON group this was the 9-15 month post-implant period.
- Intervention Pacing Features Programmed OFF: 6-month period subjects had the intervention pacing features programmed OFF. For subjects randomized to the ON-OFF group, this was the 9-15 month post-implant period. For subjects randomized to the OFF-ON group this was the 3-9 month post-implant period.
Arm/Group | Intervention Pacing Features Programmed ON | Intervention Pacing Features Programmed OFF
Number analyzed (Participants) | 222 | 222
Episodes per subject per month | 2.0 (4.8) | 1.8 (5.2)
Statistical Analysis 1: Comparison: Intervention Pacing Features Programmed ON vs Intervention Pacing Features Programmed OFF; Null Hypothesis: rate of symptomatic atrial tachycardia/atrial fibrillation episodes during periods when intervention pacing features ON is greater to or equal to the rate of symptomatic atrial tachycardia/atrial fibrillation episodes during periods where intervention pacing features were programmed OFF Alternative Hypothesis: rate of symptomatic AT/AF during periods of ON programming is less than the rate of symptomatic AT/AF during OFF programming; Test type: Superiority or Other; p = 0.629, t-test, 1 sided — P-value is from a paired t-test since each subject had the intervention pacing features turned ON and OFF in this crossover study; One-sided paired t-test with 221 degrees of freedom; Mean Difference (Final Values) = 0.1, 95% CI 1-sided [upper limit 0.5], Standard Deviation 4.8 — A mean difference greater than zero indicates an average increase in atrial fibrillation/atrial tachycardia symptomatic episodes while the intervention pacing features were programmed ON versus OFF

2. Secondary Outcome: Evaluate Subject Symptoms With the Atrial Fibrillation (AF) Symptom Checklist
Description: The AF symptom checklist (SCL) is a 16 item questionnaire measuring the frequency of 16 arrhythmia related symptoms such as tiredness/lack of energy, heart fluttering/skipping, heart racing, lightheadedness, etc. Symptom frequency is rated as never (scored as 0), rarely (scored as 1), sometimes (scored as 2), often (scored as 3), and always (scored as 4). Scores are summed across each subject and timepoint and range from 0 (no symptoms) to 64 (always symptoms). For each subject the 9 month and 15 months scores were summed respectively and ON minus OFF differences computed.
Time Frame: 6 months (per Intervention)
Population: Of the 256 randomized subjects only 211 completed the AF symptom checklist at both the 9-month and 15-month visit. Since this was a crossover study, data from both visits was required for the subject to be included in the analysis
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Intervention Pacing Features Programmed ON | Intervention Pacing Features Programmed OFF
Number analyzed (Participants) | 211 | 211
Scores on a scale | 12.0 [0 to 41] | 13.0 [0 to 41]
Statistical Analysis 1: Comparison: Intervention Pacing Features Programmed ON vs Intervention Pacing Features Programmed OFF; The null hypothesis is that the symptom frequency score does not differ between while intervention pacing features were programmed ON versus OFF. This secondary objective was not powered; Test type: Superiority or Other; p = 0.165, Wilcoxon (Mann-Whitney); P-value is from Koch's adaptation to the Wilcoxon Rank-Sum test comparing the within subject ON minus OFF differences to 0; Median Difference (Final Values) = -1.0 — A negative change means an improvement in AF symptom frequency with intervention pacing therapy programmed ON. Total possible improvement while intervention features are programmed ON is -64. Total possible worsening during ON programming is 64

3. Secondary Outcome: Time to First Cardioversion (Changing an Abnormal Heart Rhythm Into a Normal One by Using Either Medication or Electrical Shock)
Description: The dates of cardioversions attempted for atrial fibrillation (AF) since the previous study visit were collected at the 3, 9, and 15 month follow-up visits. For each randomized subject, the months to first attempted cardioversion during each randomized study period (3-9 months and 9-15 months) was determined. A repeated measures Cox proportional hazards model was used to compare the attempted cardioversion rate during periods of time where the pacing features were programmed ON versus OFF.
Time Frame: 6 months (per Intervention)
Population: All randomized subjects with follow-up during intervention pacing feature programming period.
Measure: Mean (Standard Deviation); unit: Months
Arm/Group | Intervention Pacing Features Programmed ON | Intervention Pacing Features Programmed OFF
Number analyzed (Participants) | 249 | 245
Months | 2.1 (1.7) [upper limit 1.73] | 3.3 (1.6)
Statistical Analysis 1: Comparison: Intervention Pacing Features Programmed ON vs Intervention Pacing Features Programmed OFF; Null Hypothesis: AF Cardioversion attempt rate is the same during periods of ON and OFF programming Alternative Hypothesis: AF Cardioversion attempt rate is different during periods of ON and OFF programming; Test type: Superiority or Other; p = 0.603, Regression, Cox — P-value is based on a repeated measures Cox proportional hazards model to the rate of AF cardioversion attempts between periods of ON and OFF programming; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.39 to 1.73] — Hazard Ratio compares rate of first attempted cardioversion for AF while the intervention pacing features were programmed ON versus OFF

4. Secondary Outcome: Atrial Tachycardia/Atrial Fibrillation (AT/AF) Burden
Description: AT/AF burden is defined as the sum of the duration of all atrial arrhythmias as recorded by the device divided by the device follow-up time during the programming period expressed as hours of atrial arrhythmia per day.
Time Frame: 6 months (per Intervention)
Population: Of the 256 randomized to ON-OFF or OFF-ON programming, 225 had device data necessary for computing AT/AF burden in both randomized study periods.
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | Intervention Pacing Features Programmed ON | Intervention Pacing Features Programmed OFF
Number analyzed (Participants) | 225 | 225
hours per day | 4.0 (6.8) | 4.1 (7.2)
Statistical Analysis 1: Comparison: Intervention Pacing Features Programmed ON vs Intervention Pacing Features Programmed OFF; Null Hypothesis: There is no difference in AT/AF burden during periods on ON and OFF programming Alternative Hypothesis: AT/AF burden is lower during periods of ON programming compared to periods of OFF programming; Test type: Superiority or Other; p = 0.394, Wilcoxon (Mann-Whitney) — Within each randomized subject, the ON minus OFF difference in AT/AF burden was computed. The Wilcoxon Signed-Rank test was used to determine if the ON minus OFF difference in AT/AF burden was different from zero; Median Difference (Net) = 0 — A negative median difference represents an improvement (lessening) of AT/AF burden during periods of ON versus OFF programming. A positive median difference represents an increase in AT/AF burden during ON compared to OFF programming

ADVERSE EVENTS:
Time Frame: From enrollment through the 15-month study visit
Description: Only serious adverse events when information reasonably suggested that a device had or may have caused the adverse event were collected.
Arm/Group | On-Off | Off-On | Non-Randomized Group
Serious Adverse Events (participants affected / at risk) | 7/132 | 8/124 | 4/144
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | On-Off (N=132) | Off-On (N=124) | Non-Randomized Group (N=144)
RV Lead Dislodgement (General disorders) | 1 (1) | 3 (3) | 0 (0)
Other System Effect (General disorders) | 0 (0) | 1 (1) | 1 (1)
RA Lead Dislodgement (General disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial Fibrillation (General disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation/Gastrointeritis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Device Electrical Reset (General disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Failure to Capture (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hemo/pneumothorax (General disorders) | 1 (1) | 0 (0) | 0 (0)
Other Component Failure (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pacemaker Syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pocket Erosion (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary Edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
RV and RA Lead Dislodgement (General disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The effect of ON programming was not consistent across randomized study period, violating a key assumption of the cross-over study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other